CLINICAL TRIAL: NCT01724671
Title: A Case Series of Ceftaroline-treated Patients With Infections Caused by MRSA That Are Susceptible to Ceftaroline, Compared to Vancomycin-treated Patients
Brief Title: Vancomycin Versus Ceftaroline in Patients With Infections Caused by MRSA That Are Susceptible to Ceftaroline
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CPL Associates (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Jerome Schentag, Pharm.D., CPL Associates
Other Study IDs: CPLA 6656
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: MRSA Infection; Bacteremia; ABSSSI; Pneumonia
Keywords: MRSA; Bacteremia; ABSSSI; Pneumonia; Vancomycin; Ceftaroline
MeSH Terms: conditions — Bacteremia; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — MRSA cultures obtained retrospectively from Microbiology labs if available for patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cefatroline: Investigators will retrospectively capture patient cases that have been treated for MRSA with ceftaroline. Cases will only be included if the isolate was tested against vancomycin and ceftaroline
- Vancomycin: Investigators will retrospectively capture patient cases that were been treated for MRSA with Vancomycin.

SUMMARY:
To compare the time to pathogen eradication, and the relationship to the time to clinical improvement, between ceftaroline and case-matched vancomycin treated controls in the treatment of adults with serious infections caused by Methicillin-Resistant Staphylococcus aureus (MRSA).

ELIGIBILITY:
Inclusion Criteria:

1. A positive MRSA culture, resulting from a blood or properly obtained infection site sample, with a vancomycin MIC 1.5 - 4.0 mcg/mL and ceftaroline MIC ≤1 mcg/mL.
2. The patient was treated adequately with ceftaroline or vancomycin.
3. A medical history, clinical signs and symptoms, and radiological findings consistent with infection such as pneumonia, skin and wound, intra-abdominal infection and bacteremia associated with one of those infection sites.

   Patients must have had a body temperature >38C [100.4F] or <36.1C [97F] or leukocytosis (blood leukocyte count >10,000 cells/mm3) or >10% bands, at baseline. In the case of pneumonia, chest radiographic examination that show a new or progressive infiltrate, consolidation, cavitation, or pleural effusion. Rales or dullness to percussion on physical examination of the chest, new onset of purulent sputum, or change in quantity or character of sputum. Wound redness, swelling, and/or purulence in the case of ABSSSI
4. There should be sufficient numbers of follow up cultures of the infection site and/or blood to determine whether the infecting pathogen was eradicated, and preferably the day on which the eradication occurred.

Additional inclusion criteria for patients with pneumonia:

1. Suspected or confirmed acute bacterial pneumonia due to MRSA in one of the following subgroups:

   Community-acquired bacterial pneumonia (CABP) i.e. those cases acquired outside the hospital and being admitted to the hospital for treatment of their pneumonia;

   or

   Hospital-acquired bacterial pneumonia (HABP), i.e., pneumonia that occurs 72 hours or more after admission, which was not incubating at the time of admission;

   or

   Ventilator-associated bacterial pneumonia (VABP), i.e., pneumonia that arises more than 48 hours after endotracheal intubation and ventilation;

   or

   Health Care-associated bacterial pneumonia (HCABP), which includes patients admitted from a long term care facility.
2. Pulmonary infiltration consistent with the diagnosis of pneumonia (new or progressive infiltrates, consolidation, with or without the presence of pleural effusion) documented by chest X-ray or CT within 48 hours prior to enrollment.
3. Suitable respiratory specimen (sputum/endotracheal specimen or specimen from an invasive procedure) for culture and Gram stain, with Gram-positive pathogens as the predominant organism. Average of at least 10 Gram-positive organisms per oil-immersion field in 10 fields (actual or calculated, 100x objective).

Additional inclusion criteria for patients with other infection sites:

1. In all cases of bacteremia linked to a site/source, the isolate species and susceptibility should match between blood and primary site. Typical non-pneumonia sites of infection will include complicated intra-abdominal (cIAI) and ABSSSI.
2. In contrast, bacteremic patients with IV catheter as the only source will require that the catheter was removed/replaced, and yet the patient remains culture positive for at least 24 hr after replacement of the catheter.

Exclusion Criteria

1. Age <18 years
2. Pregnant or lactating women
3. Life expectancy <3 months from underlying disease
4. Infection with Mycobacterium tuberculosis
5. Organism is not available or is not tested locally for MIC to ceftaroline or vancomycin
6. Bacteremia determined to be catheter-related with no definitive evidence of a secondary source
7. Patient is on a prior antibiotic and shows clinical improvement or negative cultures before treatment of ceftaroline (or vancomycin for control patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will retrospectively capture patient cases that have been treated for MRSA with ceftaroline, either in response to cultures or empirically with subsequent discovery of MRSA. Cases will only be included if the isolate was tested against vancomycin and ceftaroline, unless the isolate is available in the microbiology lab to send to the study coordinating center for subsequent testing of minimum inhibitory concentrations (MIC). Case matched patients treated with vancomycin will also be collected as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial Eradication | 10 days
  Time to eradication of bacteria from the infection site and/or blood in relation to time to clinical improvement. For Acute Bacterial Skin and Skin Structure Infections (ABSSSI), it is recognized that wound cultures may not be repeated often, so the focus will be on the monitoring of time to clinical resolution in conjunction with time to resolve the bacteremic phase, if bacteremia is present.

SECONDARY OUTCOMES:
Test of Cure | 10 days
  Secondary Efficacy endpoint (Cure, Failure or Indeterminate) will also be assessed at the Test of Cure, 7-10 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome J Schentag, Pharm.D., Principal Investigator — State University at Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States